CLINICAL TRIAL: NCT02584491
Title: Linking Neuroplasticity With the Outcomes of Motor Learning Based Interventions: Multi-modal Evaluation of Walking-based Training in Children and Youth With Cerebral Palsy
Brief Title: Brain Change After Fun, Athletic, Sports-skill Training (BeFAST)
Acronym: BeFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-519
Record Dates: First submitted 2015-09-17; First posted 2015-10-22 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional gait-related training (Experimental): 16 session, 6-week intensive functional gait-related training intervention based on motor learning principles that includes a motor imagery practice component.
  Interventions: Behavioral: Functional gait-related training

INTERVENTIONS:
Behavioral: Functional gait-related training — The motor learning (ML)-based functional gait-related training program is designed to improve advanced gross motor skills and athleticism. It will involve 45-min sessions twice to three times weekly over 6 weeks for a total of 16 active sessions. A maximum of 7 weeks will be permitted. Each session will consist of 35-min of active training along with a 10-min active warm-up/cool-down that incorporates ML. Scheduling flexibility will promote adherence, with a minimum one day between sessions to provide opportunity for rest. Children will be given a 3- to 5-min mental motor imagery script to practice on days when they do not have active training sessions. The total number of sessions (combined active/imagery) will be five per week.

SUMMARY:
The purpose of this study is to determine the associations between changes in neural activity and structure, advanced gross motor skills, gait characteristics, and physical activity participation following a gait-related intervention that is based on motor learning principles for ambulatory children and youth with hemiplegic and diplegic cerebral palsy. The investigators' hypothesis is that in conjunction with a program of motor learning based training, functional neuroplastic changes in the involved motor areas will be strongly associated with changes in gait and advanced gross motor skills, moderately associated with physical activity based participation changes, and will have a fair association with structural neuroplastic change.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 to17 years inclusive;
* GMFCS Level I or II;
* Able to follow testing and motor imagery instructions;
* Able to actively participate in a minimum of 45 minutes of physical activity;
* Able to independently dorsiflex both ankles;
* Able to commit to attendance of sessions two to three times weekly for six weeks.

Exclusion Criteria:

* Orthopaedic surgery within the last 9 months (muscle) or 12 months (bone);
* Botulinum toxin-A (BTX-A) injections to lower limb in the last 4 months;
* Inability to discontinue BTX-A for period of 12 weeks (during trial) due to concerns about ROM or pain;
* Severe spasticity (may be a contraindication for neuroimaging procedures);
* Seizure disorder (if not fully controlled by medication for the 12 months);
* Not prepared or unable to discontinue a regular lower limb therapy intervention during the course of the trial;
* Involved in another intervention study;
* Standard MRI contraindications (e.g., metal implants such as cochlear implant, claustrophobia).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in functional activity in lower-limb related cortical areas, assessed using functional MRI (fMRI) | 7 days pre/7 days post training intervention
Change from baseline in advanced motor skills on the Challenge Module | 7 days pre/7 days post/4-months post training intervention
  The Challenge Module is a new published measure of advanced motor skills.

SECONDARY OUTCOMES:
Change from baseline in resting state activity, assessed using resting state fMRI | 7 days pre/7 days post training intervention
Change from baseline in microstructure of brain, assessed using diffusion tensor imaging (DTI) | 7 days pre/7 days post training intervention
Change from baseline in Physical Activity self-efficacy | 7 days pre/7days post/4-months post training intervention
  Participant-report measure of Task efficacy and Barrier efficacy for physical activity.
Change from baseline in walking activity, assessed using a StepWatch accelerometer | 7 days pre/7days post/4-months post training intervention
  Participants will wear the StepWatch for 5 days.
Change from baseline in gait kinematics as measured using an electronic walkway | 7 days pre/7days post/4-months post training intervention
  Time/distance parameters of footsteps via GAITRite system.
Change from baseline in gait kinetics/kinematics as measured using 3D motion capture system | 7 days pre/7days post/4-months post training intervention
  Whole body gait analysis via Vicon motion capture and Bertec force plates.
Change from baseline in physical activity participation, as measured using the Participation and Environment Measure for Children/Youth (PEM-CY) | 7 days pre/7days post/4-months post training intervention
  Parent-report measure of participation in the home, school and community, as well as environmental factors within each setting.
Change from baseline in walk speed on the Six-minute walk test | 7 days pre/7days post/4-months post training intervention
  Standardized 6 minute walk test (with shoes, orthoses, walking devices as required) to determine distance covered (capability measure). Well-validated in pediatric CP.
Change from baseline in targeted goal abilities and satisfaction with performance as measured by the Canadian Occupational Performance Measure | 7 days pre/7days post/4-months post training intervention
  Three to five individualized walking-based activity/participation set at baseline with assessor and child/parent, and re-evaluated by child/parent at post-intervention assessments
Change from baseline in targeted goal abilities as measured by Goal Attainment Scaling (GAS) | 7 days pre/7days post/4-months post training intervention
  Three to five individualized walking-based activity/participation set at baseline with assessor and child/parent, and re-evaluated by child/parent at post-intervention assessments
Motor learning content of interventions, as assessed using the Motor Learning Strategy Rating Instrument (MLSRI) | Week 2, 4, 6
  The MLSRI is used to assess the extent to which motor learning strategies are used within an intervention session
Motor learning as evaluated using retention and transfer tests | Week 2, 4, 6
  Individualized skills will be identified to practice at every session (retention) and only at sessions 5/10/15 (transfer) to evaluate motor learning
Change from baseline in lower-limb proprioception | 7 days pre/7days post/4-months post intervention
  Lower limb joint-sense position and kinesthesia will be assessed using a semi-goniometer (protocol modified from Wingert et al, 2009)
Mental chronometry: walking | 7 days pre/7days post/4-months post intervention
  Participants will be timed while walking a 10-meter distance, and then timed while imagining walking the same distance.

OTHER OUTCOMES:
Body Pain | Completed 2 minutes before and 2 minutes after each intervention session
  Use of FACES pain scale and body diagrams to show areas of pain (musculoskeletal and other)
Intervention enjoyment, assessed using a modified version of the Physical Activity Enjoyment Scale (PACES) | Week 2, 4, 6
  Participants' enjoyment of the intervention sessions will be assessed every 2 weeks, with the questionnaire administered by a research team member not involved in intervention delivery.
Rating of exertion, assessed using Pictoral Children's Effort Rating Table (PCERT) | Completed at 22 minutes (mid-point) and at 43-minutes (2-minutes before end) of each intervention session
  Children will be asked to complete PCERT at mid-point of each session, and 2 minutes before session completion
Heart Rate | Assessed at 4 time points per session: 1 min before start of session, at 22 minutes (mid-point), at 43-minutes (2-min before end), and at 45-minutes (end) of each session.
  Heart rate will be monitored by treating kinesiologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hilderley AJ, Wright FV, Taylor MJ, Chen JL, Fehlings D. Functional Neuroplasticity and Motor Skill Change Following Gross Motor Interventions for Children With Diplegic Cerebral Palsy. Neurorehabil Neural Repair. 2023 Jan;37(1):16-26. doi: 10.1177/15459683221143503. Epub 2022 Dec 15. PMID 36524254